CLINICAL TRIAL: NCT06962800
Title: An Open-Label, Multicenter, Randomized Phase 3 Study Evaluating the Efficacy and Safety of Felzartamab in Participants With Primary Membranous Nephropathy (PMN) [PROMINENT]
Brief Title: A Study to Learn More About the Effects and Safety of Felzartamab Infusions in Adults With Primary Membranous Nephropathy (PMN)
Acronym: PROMINENT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 299PN301; 2024-519232-16-00 (Other: EU CT Number)
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Primary Membranous Nephropathy
MeSH Terms: interventions — felzartamab; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Open-Label Treatment Phase (Experimental): Participants will receive several intravenous (IV) doses of felzartamab or oral tacrolimus in the Open-Label Treatment Phase.
  Interventions: Drug: Felzartamab; Drug: Tacrolimus
- Non-Responder Treatment Phase (Experimental): Participants initially randomized to felzartamab or tacrolimus who meet rescue criteria may receive regional standard of care immunosuppressive therapy (IST) per Investigator discretion or several IV doses of felzartamab, respectively, in the Non-Responder Treatment Phase.
  Interventions: Drug: Felzartamab; Drug: Standard of Care IST

INTERVENTIONS:
Drug: Felzartamab — Administered intravenously
  Other Names: MOR202, MOR03087, TJ202, BIIB148, HIB202
Drug: Tacrolimus — Administered orally
  Arms: Open-Label Treatment Phase
Drug: Standard of Care IST — Administered intravenously and orally
  Arms: Non-Responder Treatment Phase

SUMMARY:
In this study, researchers will learn more about the use of felzartamab in participants with primary membranous nephropathy, also known as PMN. In people with PMN, autoantibodies build up in the glomeruli of the kidney. Antibodies are proteins that help the body fight off infection. An autoantibody is a type of antibody that mistakenly targets and attacks the body's own tissues. Glomeruli are the filters of the kidney that remove waste and extra fluid from the body. In PMN, the build-up of autoantibodies in the glomeruli causes damage to the kidneys.

Kidney damage can lead to too much protein and blood leaking into the urine. High levels of protein in the urine, called proteinuria, are common in people with PMN. Symptoms of PMN can include swelling in the legs and body, tiredness, and high blood pressure. If left untreated, PMN can eventually lead to kidney failure.

In this study, researchers will learn more about how a study drug called felzartamab affects people with PMN. Felzartamab is a monoclonal antibody, which means it is an antibody made in a laboratory. Felzartamab can target immune cells that produce autoantibodies, helping to lower their buildup in the kidneys. The main goal of this study is to compare how felzartamab works compared to a drug called tacrolimus. Tacrolimus is another drug given to people with PMN and kidney disease.

The main question that researchers want to answer is:

* How many participants achieve a complete response after 104 weeks of treatment?
* A complete response means that their urine protein levels decrease to a low level and their kidney function remains stable.

Researchers will also learn about:

* How long it takes before the participants' disease gets worse
* How long the participants' urine protein levels stay low
* How many participants develop antibodies against felzartamab in the blood?
* How many participants achieve a complete response after 76 weeks of treatment
* How many participants have medical problems during the study
* How felzartamab is processed by the body
* How felzartamab affects participants' tiredness and overall physical health

The study will be done as follows:

* Participants will be screened to check if they can join the study. This may take up to 42 days.
* Participants will be randomized to receive either felzartamab as intravenous (IV) infusions or tacrolimus, taken orally as tablets.
* If participants have worsening kidney function or worsening proteinuria, or if their PMN relapses, or if they show no signs of improvement in their PMN, they will have a chance to receive rescue treatment.
* If a participant stops treatment early, there will be follow-up visits every 12 weeks until they reach Week 104.
* In total, participants will have up to 23 study visits. Participants who do not need rescue treatment will stay in the study for up to 104 weeks. Participants who need rescue treatment will stay in the study for up to 156 weeks.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the efficacy of felzartamab compared to tacrolimus in participants with PMN in achieving complete remission (CR) of proteinuria. The secondary objectives of the study are to evaluate the efficacy of felzartamab through additional clinical endpoints and timepoints, to assess the impact of felzartamab on serum anti-phospholipase A2 receptor (PLA2R) antibodies and patient-reported outcomes, and to assess the safety, pharmacokinetics (PK) and immunogenicity of felzartamab.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with PMN in need of IST according to the Investigator's clinical judgment. The diagnosis of PMN must be documented with the presence of nephrotic syndrome, and hypoalbuminemia, and confirmed with a kidney biopsy either during Screening or within 5 years of signing the informed consent form (ICF) [see kidney biopsy exception below for participants positive for anti-PLA2R antibodies]. For these participants, the biopsy report with redacted protected health information must be available to be reviewed by the Sponsor or an independent nephropathologist. If the participant requires a kidney biopsy during Screening, medical monitor approval must be obtained and all other eligibility criteria should be reviewed to ensure that the participant is otherwise eligible prior to performing the kidney biopsy.

  a. Kidney biopsy exception for anti-PLA2R antibody positive participants: Participants who are positive for anti-PLA2R antibodies and have not had a kidney biopsy performed within 5 years of signing the ICF, may be eligible for the study without undergoing a kidney biopsy based on medical monitor review confirming normal estimated glomerular filtration rate (eGFR), presence of nephrotic syndrome, hypoalbuminemia, positive anti-PLA2R antibody test (defined as an anti-PLA2R antibody titer > 20 RU/mL), and documentation provided by the Investigator that the work-up for secondary causes of membranous nephropathy (MN) was negative with no identifiable secondary causes.
* Meets one of the following:

  1. Newly diagnosed PMN, defined as having never received IST for PMN in the past.
  2. Relapsed PMN, defined as documented achievement of CR or partial remission (PR) after treatment with an IST for PMN followed by reappearance of nephrotic range proteinuria (urine protein to creatinine ratio [UPCR] ≥ 3.0 gram per gram [g/g] from a 24-hour urine collection or proteinuria ≥ 3.5 gram per 24 hour [g/24 h]).
* Participants must be on the maximally approved dose or maximally tolerated dose of angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) for at least 3 months prior to Screening. Participants not on the maximally approved dose of renin-angiotensin-aldosterone system (RAAS) inhibition may be enrolled provided there is documented intolerance to maximal RAAS inhibition (e.g., angioedema, development of postural hypotension, lightheadedness, hyperkalemia, etc).
* A UPCR of ≥ 3.0 g/g (as determined by a 24-hour urine collection) or total proteinuria ≥ 3.5 g/24 h (as determined by a 24-hour urine collection) at Screening after best supportive care for at least 3 months prior to signing the ICF.

Key Exclusion Criteria:

* Secondary cause of MN (e.g., malignancies, medications, systemic lupus erythematosus [SLE], hepatitis B, hepatitis C, etc).
* Severe renal impairment defined as an eGFR ≤ 30 mL/min/1.73m^2 at Screening or including the need for dialysis or renal replacement therapy.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2028-12-29 (Estimated); Study Completion 2029-03-29 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Complete Remission (CR) at Week 104 | Week 104

SECONDARY OUTCOMES:
Percentage of Participants who Achieve Overall Remission (OR), Defined as CR or Partial Remission (PR) at Week 104 | Week 104
Percentage of Participants who Achieve CR at Week 76 | Week 76
Duration of CR | Baseline up to week 156
Percentage of Participants With a Baseline Anti-Phospholipase A2 Receptor (PLA2R) Autoantibody Titer Greater Than 50 Relative Unit per Milliliter (RU/mL) who Achieve an OR at Week 76 and at Week 104 | Weeks 76 and 104
Time to Disease Worsening | Baseline up to week 156
Time to a Sustained Reduction in eGFR of ≥ 30% From Baseline | Baseline up to week 104
Absolute Change in Anti-PLA2R Autoantibody Titer in Participants Positive for Anti-PLA2R at Baseline | Baseline up to week 156
Change From Baseline in the Patient Reported Outcome Measurement Information System (PROMIS) Fatigue Scale at Week 104 | Week 104
Change From Baseline in PROMIS Global Assessment of Physical Health Scale at Week 104 | Week 104
Number of Participants With Treatment Emergent Adverse Event (TEAE), Serious Adverse Event (SAE) and Adverse Events of Special Interest (AESIs) | From first dose of study drug up to end of follow-up (up to week 156)
Felzartamab Serum Concentrations Over Time | Predose and at multiple timepoints post dose up to week 156
Number of Participants With Anti-Drug Antibodies (ADAs) Against Felzartamab | Predose and at multiple timepoints post dose up to week 156

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (59):
- United States (10):
  - Apogee Clinical Research, LLC, Huntsville, Alabama
  - The Nephrology Group, Inc. - Fresno, Fresno, California
  - Academic Medical Research Institute, Los Angeles, California
  - Henry Ford Hospital- A-Basement Research Pharmacy, Detroit, Michigan
  - Elixia Health - Michigan Kidney Consultants, LLC - Elixia - PPDS, Pontiac, Michigan
  - James J Peters Veterans Administration Medical Center - NAVREF - PPDS, The Bronx, New York
  - ECU Physicians Nephrology and Hypertension, Greenville, North Carolina
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - Nephrotex Research Group, Dallas, Texas
  - University of Texas Medical Branch, League City, Texas
- Argentina (5):
  - Organización Médica de Investigación, Buenos Aires
  - CINME S.A. - Centro de Investigaciones Metabólicas, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Clínica Privada Vélez Sarsfield, Córdoba
- Australia (4):
  - Concord Hospital, Concord, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Townsville Hospital, Douglas, Queensland
  - Griffith University Clinical Trial Unit, Southport, Queensland
- Brazil (4):
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul (PUCRS), Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto da Universidade de Sao Paulo, Ribeirão Preto, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto Hospital de Base - PPDS, São José do Rio Preto, São Paulo
  - Centro de Pesquisa Clínica de Nefrologia do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
- China (14):
  - Fu Yang People's Hospital - South Campus, Fuyang, Anhui
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital - Changqiao Campus, Xichengqu Beijing, Beijing Municipality
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Second Hospital of Hebei Medical University - Main, Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The First Affiliated Hospital of Henan Science and Technology University - Jinghua Campus, Luoyang, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Yueyang People Hospital, Yueyang, Hunan
  - Qilu Hospital of Shandong University, Jinan, Shandong
- Japan (8):
  - National Hospital Organization Chiba Medical Center Chibahigashi National Hospital, Chia-shi, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaidô
  - Kagawa University Hospital, Kita-Gun Uchiko-Cho, Kagawa-ken
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - University of Miyazaki Hospital, Miyazaki, Miyazaki
  - Niigata University Medical ＆ Dental Hospital, Niigata, Niigata
  - Social Medical Corporation Yuuaikai Yuuai Medical Center, Tomigusuku-Shi, Okinawa
  - Japanese Red Cross Musashino Hospital, Musashino-shi, Tokyo
- Malaysia (2):
  - Hospital Raja Permaisuri Bainun, Perak, Pahang
  - Hospital Canselor Tuanku Muhriz UKM, Cheras, WilayahPersekutuan KualaLumpur
- South Korea (5):
  - Ajou University Hospital, Suwon, Gyeonggido
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Inje University Haeundae Paik Hospital, Busan
  - Hanyang University Seoul Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
- Taiwan (7):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - MacKay Memorial Hospital, Taipei
  - Taipei Medical University Hospital - PPDS, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/